CLINICAL TRIAL: NCT06125847
Title: A Clinical Study for the Safety and Efficacy of Intravenous Infusion of NGGT006 in Treatment of Homozygous Familial Hypercholesterolemia With LDLR Mutations
Brief Title: NGGT006 Gene Therapy for Homozygous Familial Hypercholesterolemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NGGT006-P-2301
Record Dates: First submitted 2023-10-30; First posted 2023-11-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-09

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: Homozygous familial hypercholesterolemia; Gene therapy; Low-density lipoprotein cholesterol
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NGGT006 (Experimental): 4 doses of NGGT006 will be administered according to the principle of dose escalation
  Interventions: Genetic: NGGT006

INTERVENTIONS:
Genetic: NGGT006 — Single intravenous infusion of NGGT006 at dose 1 (7.5e12vg/kg), dose 2 (1.5e13vg/kg) , dose 3 (3e13vg/kg) and dose 4 (4e13vg/kg).

SUMMARY:
This is an early phase 1, open-label, single-center, dose-escalation, pilot trial to evaluate the safety and efficacy of an intravenous infusion of NGGT006 in homozygous familial hypercholesterolemia (HoFH) patients with LDLR mutations. NGGT006 is an adeno-associated viral (AAV) vector carrying codon-optimized human LDLR gene, driving the expression of LDLR protein with normal function and promoting the clearance of low-density lipoprotein cholesterol (LDL-C).

DETAILED DESCRIPTION:
Homozygous familial hypercholesterolemia (HoFH) is a rare inherited disorder of lipoprotein metabolism, characterized by extreme elevations in low-density lipoprotein cholesterol (LDL-C) and leading to early onset of severe coronary artery disease. This is an early phase 1, open-label, single-center, dose-escalation, pilot trial to evaluate the safety and efficacy of a single intravenous infusion of NGGT006 in HoFH patients with LDLR mutations. NGGT006 is an adeno-associated viral (AAV) vector carrying codon-optimized human LDLR gene, driving the expression of LDLR protein with normal function and promoting the clearance of low-density lipoprotein cholesterol (LDL-C). 4-15 subjects will be enrolled and divided into 4 groups according to the principle of dose escalation, respectively administered intravenous infusion of NGGT006 at dose group 1 (7.5e12vg/kg), dose group 2 (1.5e13vg/kg) , dose group 3 (3e13vg/kg) and dose group 4 (4e13vg/kg). The researcher is allowed to extend 0-3 patients. All subjects will undergo 52 weeks of treatment observation and further 260 weeks of long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign informed consent form;
* Male or female, 12 ≤ age ≤ 55 years (first patient≥ 18 years), diagnosed as homozygous familial hypercholesterolemia with genetic confirmation of two mutant alleles of the LDL receptor (LDLR) gene;
* AAV8 neutralizing antibodies can be negative or reduced to negative levels through methods such as plasma exchange.
* Untreated LDL-C ≥10 mmol/L (386mg/ dL) or treated LDL-C ≥7 mmol/L (270mg/ dL) together with cutaneous or tendon xanthoma before age 18 years;
* Had been on stable medication for ≥30 days if receiving lipid-lowering therapy (or ≥60 days if receiving alirocumab or evolocumab) prior to screening and not scheduled for addition of new drugs or dose adjustments during the study;
* Agreed to follow a low-fat diet and comply with all study procedures;
* Agreed to maintain a similar exercise volume and intensity to baseline during the study period;
* Agreed to maintain good lifestyle habits;
* No history of alcohol abuse or alcohol dependence (diagnosed as F10 in ICD-10 code);
* No sexual activity for 14 days prior to administration and negative serum pregnancy test in female participants;
* Participants of childbearing potential agreed to use highly effective contraception for at least 365 days from administration of NGGT006;
* No plan of stent implantation within 3 months.

Exclusion Criteria:

* Positive for hepatitis B surface antigen, hepatitis C, human immunodeficiency virus (HIV) or syphilis test;
* Clinically significant abnormalities in liver function test: alanine aminotransferase (ALT) ≥2 × upper limit of normal (ULN) and/or aspartate aminotransferase (AST) ≥2 × ULN;
* Baseline blood pressure ≥160/100 mmHg (1 repeat measurement is allowed);
* Uncontrolled myocardial infarction or heart failure, or had surgery plan within 1 year;
* Diabetes diagnosed within 3 months or with poor control (HbA1c ≥9%);
* Acute or chronic kidney failure;
* Hemoglobin (Hb) ≥120g/L (male), Hb ≥110 (female);
* Abnormal platelet counts or morphology;
* History or laboratory tests suggestive of thrombosis;
* Had contraindications to glucocorticoid (e.g., epilepsy, severe schizophrenia, active peptic ulcer);
* Life expectancy less than 1 year;
* With malignant tumors;
* Liver fibrosis or liver cancer;
* Previous gene therapy treatment;
* Hypersensitivity to AAV or cortisone or immunosuppressants (sirolimus, rituximab, tacrolimus);
* Participation in any other clinical trial within 3 months;
* History of stent implantation within 1 month or myocardial infarction within 3 months;
* Breastfeeding females;
* Any other condition that may not be appropriate for the study in the opinion of the Investigator.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-29 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (AE) and serious adverse events (SAE) | 52 weeks
  Incidence of AE and SAE, as assessed by physical examinations, clinical laboratory parameters and adverse event reporting
Absolute change and percent change in LDL-C | 52 weeks
  Change in LDL-C concentration from baseline to week 52

SECONDARY OUTCOMES:
Absolute change and percent change in apoB | 52 weeks
  Change in lipid concentrations from baseline to week 52
Absolute change and percent change in TC | 52 weeks
  Change in lipid concentrations from baseline to week 52
Absolute change and percent change in HDL-C | 52 weeks
  Change in lipid concentrations from baseline to week 52
Absolute change and percent change in TG | 52 weeks
  Change in lipid concentrations from baseline to week 52
Absolute change and percent change in Lp(a) | 52 weeks
  Change in lipid concentrations from baseline to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Zuyi Yuan, M.D., Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No